CLINICAL TRIAL: NCT01858246
Title: A Randomised Controlled Trial Comparing Bone Anchored Hearing Aid With Bonebridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ninewells Hospital (Other)
Responsible Party: Principal Investigator, Stephen Jones, Consultant ENT Surgeon, Ninewells Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJPSMH01
Record Dates: First submitted 2013-05-15; First posted 2013-05-21 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Hearing Loss, Conductive; Bone Conduction Deafness
Keywords: Hearing Loss, Conductive; Bone Conduction; bone conduction thresholds better than 45 dBHL
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bonebridge (Active Comparator): Implantation with a Bonebridge
  Interventions: Device: Bonebridge
- Bone Anchored Hearing Aid (Active Comparator): Implantation with a Bone Anchored Hearing Aid
  Interventions: Device: Bone Anchored Hearing Aid

INTERVENTIONS:
Device: Bonebridge
  Arms: Bonebridge
Device: Bone Anchored Hearing Aid
  Arms: Bone Anchored Hearing Aid

SUMMARY:
The Bonebridge is a new bone conducting implantable hearing aid. The investigators plan to randomize patients to receive either the Bonebridge or a conventional bone conducting hearing device. The investigators will then compare the surgical and audiological outcomes of the two groups.

DETAILED DESCRIPTION:
The new Bonebridge fully implanted, except for an external sound processor. It does not have any percutaneous parts like the Bone Anchored Hearing Aid. The investigators believe that this may improve wound healing and reduce problems with wound infection and skin overgrowth seen in Bone Anchored Hearing Aids.

There may also be audiological improvements by the use of the Bonebridge as the physical separation of the vibrating part from the sound processor should reduce feedback. The company also claims other audiological improvements in the Bonebridge.

The investigators wish to demonstrate whether this is actually the case by performing a study directly comparing the outcomes of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Conductive Hearing Loss within criteria for Bonebridge
* Adults

Exclusion Criteria:

* Children
* Pregnancy

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Speech audiogram result at 6 months after switch on at 60 dBA in quiet using AB word lists | Up to 1 year post-operatively
  We will record and compare the standard speech audiometry results at a specific sound level in order to make a direct comparison of devices

SECONDARY OUTCOMES:
Speech audiogram result at 60 dB A in noise using AB word lists | Up to 1 year after implantation
  The speech audiogram will also be carried out in noise to demonstrate whether one device gives an appreciable advantage over another with respect to understanding in noise compared to silence.
Patient reported outcome data | Up to 1 year following implantation
  Patients will be asked to complete the Glasgow Benefit Inventory (GBI) and Hearing Device Satisfaction Scale (HDSS) questionnaires
Time from surgery to device switch-on | Up to 3 months
  The time (measured in days) will be recorded from the date of implantation to the date of its switch-on.
Number of patient episodes required during study period | 1 year from implantation
Time to complete wound healing | Up to 3 months from implantation
  Measured in days, as judged subjectively by ENT medical and nursing staff

CONTACTS AND LOCATIONS:
Overall Officials: Stephen EM Jones, Principal Investigator — NHS Tayside
Locations (1):
- Ninewells Hospital and Medical School, Dundee, United Kingdom